CLINICAL TRIAL: NCT04503447
Title: Severe Acute Respiratory Syndrome Coronavirus (CoV) 2 (SARS-CoV-2) Seroprevalence Study in Institute of Tropical Medicine (ITM) Staff
Brief Title: COVID-19 Seroprevalence Study in ITM Staff
Acronym: CovAb
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: SARSCOV2SEROPREVALENCEITMSTAFF
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: humans; COVID-19; pandemics; SARS virus; cross-sectional studies; seroepidemiological studies; Belgium; risk factors; seroprevalence
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Belgium, the corona virus disease 2019 (COVID-19) epidemic is in the growing phase of its second wave.

The Belgian crisis cell is balancing between allowing the economy to recover and minimize the disease spread. To decide which containment measures should be maintained, reinstalled or suspended, information on what proportion of people has been infected and on possible risk factors for virus transmission can be helpful.

This study will be conducted on staff members of the ITM. All staff members will be invited to participate. Participants will be asked to have a blood sample drawn for detections of antibodies against SARS-CoV-2 (using one of these two commercial assays: Anti-SARS-CoV-2 ELISA (EUROIMMUN) or WANTAI SARS-CoV-2 Ab ELISA (WANTAI SARS-CoV-2 Diagnostics)) and to complete a questionnaire about their exposure, both within and outside the ITM, to the SARS-CoV-2, and about their health and symptoms. The primary objective is to estimate the occurrence rate of anti-SARS-CoV-2 antibodies or seroprevalence in ITM staff. Secondary objective is to estimate the SARS-CoV-2 seroprevalence in ITM staff member groups, stratified by variables obtained through the questionnaire, such as age, gender, symptoms, exposure to COVID-19 patients/samples, comorbidities, adherence to containment measures.

DETAILED DESCRIPTION:
The study is observational and will be conducted on ITM staff members. All members will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Be an active ITM staff member
* Be willing and able to complete the questionnaire
* Be willing and able to provide informed consent

Exclusion Criteria:

* Doctor of Philosophy (PhD) students, Master students and interns of the ITM

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Active ITM staff members
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 seroprevalence ITM staff | Sample is drawn once, within 7 days after recruitment
  The proportion of participating ITM staff members with detectable SARS-CoV-2 antibodies

SECONDARY OUTCOMES:
SARS-CoV-2 seroprevalence in ITM staff, stratified by variables | Questionnaire is completed once, at recruitment
  SARS-CoV-2 seroprevalence in ITM staff members stratified by variables obtained through the questionnaire, such as age, gender, symptoms, exposure to COVID-19 patients/samples, comorbidities, adherence to containment measures.

OTHER OUTCOMES:
Risk or protective factors for SARS-CoV-2 seropositivity | Questionnaire is completed once, at recruitment
  To identify factors that are associated with an elevated or reduced risk of seropositivity in ITM staff and the Belgian working population in general.

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Van Esbroeck, MD, Principal Investigator — Institute of Tropical Medicine, Belgium
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Study population being only ITM staff members, individual participant data (IPD) cannot be shared due to privacy reasons